CLINICAL TRIAL: NCT03326531
Title: Slipped Capital Femoral Epiphysis; Changes in Gait, Balance and Muscle Activity Patterns in Patients Treated With Single Screw in Situ Fixation Investigated Using Computer Assisted Rehabilitation ENvironment (CAREN)
Brief Title: "Gait and Balance in Patients With SCFE"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL56402.068.16
Record Dates: First submitted 2017-09-27; First posted 2017-10-31 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-09

CONDITIONS: Slipped Capital Femoral Epiphyses
MeSH Terms: conditions — Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable for this study — Not applicable for this study

SUMMARY:
Slipped Capital Femoral Epiphysis (SCFE) treated with one screw in situ fixation results in an altered gait. It is thought that the protraction of the pelvis at the affected side, seen in patients with unilateral stable SCFE, is a compensatory mechanism to reduce out-toeing and thereby improve foot positioning during gait. This study will evaluate this hypothesis since only a few studies are conducted evaluating gait in treated SCFE. It is also thought that this pathology results in an impaired balance. Computer Assisted Rehabilitation Environment (CAREN) will be used to investigate these two questions.

DETAILED DESCRIPTION:
Rationale: Slipped Capital Femoral Epiphysis (SCFE) treated with one screw in situ fixation results in an altered gait. It is thought that the protraction of the pelvis at the affected side, seen in patients with unilateral stable SCFE, is a compensatory mechanism to reduce out-toeing and thereby improve foot positioning to restores the gait patterns towards a 'normal gait pattern. The goal of this study is to investigate this hypothesis since only a few studies are conducted evaluating gait in treated SCFE. It is also thought that this pathology results in an impaired balance. Computer Assisted Rehabilitation Environment (CAREN) will be used.

Objective: The primary objective of this study is to investigate whether protraction of the pelvis at the affected side is a compensatory mechanism to reduce out-toeing and thereby improve foot positioning and restores the gait pattern towards a 'normal' gait pattern in patients with unilateral stable SCFE, treated with single screw in situ fixation. Dynamic postural balance will be analysed as well since an altered, waddling gait, is observed in patients with treated SCFE. In addition, activity patterns of lower limb muscles will also be evaluated using surface electromyography. Kinematic and EMG data of patients will be compared with data of healthy controls with no gait pathology in order to investigate these objectives.

Secondary objectives are the evaluation of clinical outcomes and spatiotemporal parameters in these patients compared to healthy controls.

Study design: a comparative cross-sectional case-control study.

Study population: Children and adolescents with stable SCFE managed with single screw in situ fixation and an age, gender and BMI matched healthy controls without gait pathology. Patients were excluded if major complications occurred due to in situ fixation, if they had revision surgery or had additional pathology leading to gait alterations. In addition, patients are required to walk without walking aid for at least 30 minutes.

Main study parameters/endpoints: Kinematic data will be studied at pelvis, hip, knee and ankle level. Margins of stability will be calculated to analyse dynamic postural balance. In addition, lower extremity muscle activation patterns of SCFE patients will be recorded to assess muscle activation pattern during gait. Correlations between the severity of initial slip and the clinical outcome after treatment will be evaluated.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk of CAREN based gait analysis is negligible. A safety harness provides protection against falling. It will avoid subject falling on or off the treadmill while performing training. The safety harness is secured with a life line to the ceiling. The burden of the children or adolescents is minimal. Participants will visit the MUMC+ once, where questionnaires (Hip Injury Osteoarthritis Outcome Score, SF-36 questionnaires, Borg CR10 Score and NRS score) physical examination and gait analysis will be performed. The whole session will take 2 hours. Due to the nature of the study, this study can only be done using this specific patient group.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 8 and 21 years.
* Unilateral stable SCFE, with clinical and radiological confirmation and lateral slip angles ranging from mild (LSA <30°), moderate (LSA 30°-50°) to severe (LSA >50°) based on the method of Southwick.
* Treatment of the slip with single screw in situ fixation in the last ten years, with no evidence of major complications related to the procedure like chondrolysis, avascular necrosis and infection or slip progression. Follow up at our institution for at least one year.
* Ability to walk 30 minutes without aid.
* Is able to speak, read and write the Dutch language

Exclusion Criteria:

* Clinical or radiological evidence of a contralateral slip or an endocrinopathy as underlying cause of SCFE.
* Revision surgery.
* Other pathology leading to gait alterations.

Ages: 8 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: We expect that no major deviations in gait pattern occur later than 6 months after the intervention and therefore, a stable gait pattern is presented 6 months postoperatively. This expectation is made based on clinical experience, in which gait is often affected during these first 6 months after the intervention due to pain, a long non-weightbearing period of the leg in the postoperative phase and rehabilitation. After these six months no further deviations in gait pattern were expected and a stable, compensating gait pattern is observed and patients will be analysed between 6 months till 10 years postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Joint range of motion | During an entire gait cycle while walking on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Range of motion (i.e. maximal angle minus minimal angle in degrees) of the pelvis, hip, knee and ankle of the affected and unaffected side in degrees.

SECONDARY OUTCOMES:
Absolute joint angles | During an entire gait cycle while walking on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Absolute joint angles of the pelvis, hip, knee and ankle of both the affected and unaffected side in degrees.
Margins of Stability | During an entire gait cycle while walking on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Margins of Stability is a measure to describe balance during gait
Muscle activation patterns | During an entire gait cycle while walking on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Muscle activation patterns of lower limb muscles will be recorded during gait by using EMG
Gait velocity | During an entire gait cycle while walking on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Gait velocity (in m/sec)
Hip Injury and Osteoarthritis Outcome Score | One minute before the start of the test on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Scoring system to assess general outcome after hip surgery
SF-36 questionnaire | One minute before the start of the test on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Scoring system to assess quality of life after hip surgery
Borg CR10 scale | One minute before the test on the CAREN system and one minute after the last gait cycle walked on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Scoring system to assess the severity of tiredness during the test
NRS/VAS score | One minute before the test on the CAREN system and one minute after the last gait cycle walked on the CAREN system during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Scoring system to assess pain during the test
Radiological outcome | Assessed during the only study visit moment (e.g. 6 months till 10 years after surgery).
  The Southwick Angle is used to assess the severity of initial slip
Cadence (in steps/min) | During the entire gait cycle while walking on the CAREN system, during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Cadance (in steps/min)
Step width (in cm) and stride length (in cm) | During the entire gait cycle while walking on the CAREN system, during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Step width and stride length (in cm)
Time of the gait cycle spent in stance (in seconds) | During the entire gait cycle while walking on the CAREN system, during the only study visit moment (e.g. 6 months till 10 years after surgery).
  Stance phase (in seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No